CLINICAL TRIAL: NCT01677741
Title: Phase I/IIa, 2-Part, Multi-Center, Single-Arm, Open-Label Study to Determine the Safety, Tolerability and Pharmacokinetics of Oral Dabrafenib in Children and Adolescent Subjects With Advanced BRAF V600-Mutation Positive Solid Tumors
Brief Title: A Study to Determine Safety, Tolerability and Pharmacokinetics of Oral Dabrafenib In Children and Adolescent Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116013; 2012-001499-12 (EudraCT Number); CDRB436A2102 (Other: Novartis)
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Neoplasms, Brain
Keywords: Children and Adolescents; BRAF; dabrafenib; dose escalation; BRF116013; V600-mutation positive; BRF
MeSH Terms: conditions — Brain Neoplasms | interventions — dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Dabrafenib treatment (Experimental): Three subjects will receive a single dose of 3 mg/kg dabrafenib on Day 1 and repeat dose will begin from Day 2, evenly divided in two daily doses. Once all 3 subjects have been fully evaluated for the first 28 days (including Day 15 PK) and no DLTs are observed, a next subject will be enrolled at the next higher dose levels (i.e., dose escalation to 3.75 mg/kg [+1] and may be further to 4.5 mg/kg [+2] and so on). If all 3 subjects have not been fully evaluated for the first 28 days or 1 DLT occurred, the fourth subject will be enrolled at the same dose level. If 2 or more DLTs are observed, the next subject will be enrolled at the next lower dose level (i.e., de-escalated to 2.25 mg/kg [-1] and may be further to 1.5 mg/kg [-2]). Similarly, the process is repeated for the fifth and sixth subjects in a cohort. All subjects will receive treatment till end of study.
  Interventions: Drug: Dabrafenib
- Part 2: Cohort 1 Low-Grade Gliomas with BRAF V600 mutations (Experimental): Subjects with low-grade gliomas with BRAF V600 mutations will receive the single selected final dose (based on MTD and the age of the subjects) from Part 1 on Day 1. Repeat dosing will begin from Day 2, twice daily till end of study.
  Interventions: Drug: Dabrafenib
- Part 2: Cohort 2 High-Grade Gliomas with BRAF V600 mutations (Experimental): Subjects with high-grade gliomas with BRAF V600 mutations will receive the single selected final dose (based on MTD and the age of the subjects) from Part 1 on Day 1. Repeat dosing will begin from Day 2, twice daily till end of study.
  Interventions: Drug: Dabrafenib
- Part 2: Cohort 3 LCH with BRAF V600 mutations (Experimental): Subjects with LCH with BRAF V600 mutations will receive the single selected final dose (based on MTD and the age of the subjects) from Part 1 on Day 1. Repeat dosing will begin from Day 2, twice daily till end of study.
  Interventions: Drug: Dabrafenib
- Part 2: Cohort 4 Melanoma and PTC with BRAF V600 mutations (Experimental): Subjects with other tumors with BRAF V600 mutations will receive the single selected final dose (based on MTD and the age of the subjects) from Part 1 on Day 1. Repeat dosing will begin from Day 2, twice daily till end of study.
  Interventions: Drug: Dabrafenib

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib is available as 50 mg or 75 mg capsules and as oral suspension (10 mg/mL for subjects unable to swallow capsules). Dabrafenib (either formulation) will be administered orally as a single dose on Day 1 and twice daily from Day 2, based on weight at the appropriate study dose level.
  Other Names: DRB436

SUMMARY:
This was a 2-part, Phase I/IIa, multi-center, open label, study in pediatric and adolescent patients with advanced BRAF V600 mutation-positive solid tumors. Part 1 was a dose escalation study in patients with any BRAF V600 mutation-positive solid tumor using a modified Rolling 6 Design (RSD). Part 2 was an expansion study to further evaluate the safety, tolerability, and clinical activity of dabrafenib in 4 tumor-specific pediatric populations. Patients participated in only either part 1 or part 2 of the study.

DETAILED DESCRIPTION:
Part 1 was a dose escalation study in subjects with any BRAF V600 mutation-positive solid tumor, designed to optimize efficiency of enrollment, minimize the number of subjects being treated at potentially sub-efficacious dose levels, and incorporating the evolving pharmacokinetic, safety and efficacy data from the adult development program. Dose escalation part of the study was to determine the maximum tolerated dose (MTD) and recommend the dose for phase 2 studies (RP2D). An MTD has not been identified for dabrafenib in the adult population. This does not preclude the identification of an MTD in the pediatric population. Modified RSD was employed to determine the MTD. Part 1 used dual criteria of dose limiting toxicity (DLT) and observed dabrafenib exposures to make decisions to advance to the next dose level. Target exposure criteria based on adults treated at the approved adult dose of 300 mg (150 mg given BID) were observed in this study before meeting criteria for stopping dose escalation due to observations of DLTs, and served as the criteria for determining the RP2D for dabrafenib in pediatric subjects. Thus, MTD has not been established in pediatric population, similar to the previous dose finding efforts in adult subjects.

Part 2 was a tumor specific expansion study to further evaluate the safety/tolerability profile and to discover possible clinical efficacy of dabrafenib in 4 tumor-specific pediatric populations known to have BRAFV600 activation: high grade glioma (HGG), low grade glioma (LGG), Langerhans cell histiocytosis (LCH), miscellaneous tumors including melanoma and papillary thyroid carcinoma (Other). The exposures for subjects dosed on the basis of weight were also evaluated by age categories.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent - a signed informed consent and/or assent (as age appropriate) will be obtained according to institutional guidelines.
* Male or female >=12 months and <18 years of age at the time of signing the informed consent form.
* Recurrent disease, refractory disease, or progressive disease after having received at least one standard therapy for their disease. Note: Subjects with metastatic (and surgically unresectable) melanoma can be enrolled for first-line treatment; Melanoma subjects with CNS involvement may be enrolled.
* At least one evaluable lesion.
* BRAF V600 mutation-positive tumor as confirmed in a Clinical Laboratory Improvement Amendments (CLIA)-approved laboratory or equivalent (the local BRAF testing may be subject to subsequent verification by centralized testing; centralized testing can confirm V600E and V600K mutations only).
* Performance score of >=50% according to the Karnofsky/Lansky performance status scale (subjects with a performance status of <=50% can be enrolled if the subject's confinement to bed and inability to carry out activities is due solely to cancer-related pain, as assessed by the investigator).
* Females of child-bearing potential (with negative serum pregnancy test within 7 days prior to the first dose of study medication) must be willing to practice acceptable methods of birth control .
* Sexually active males, who do not agree to abstinence, must be willing to use a condom during intercourse while taking the study drug, and for 16 weeks after stopping treatment and should not father a child in this period.
* Must have adequate organ function as defined by the following values: Adequate bone marrow function defined as-absolute neutrophil count (ANC) >=1000/ microliter (µL), hemoglobin >=8.0 grams (g)/ deciliter (dL) (may receive red blood cell transfusions), platelets >=75,000/µL (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment).
* Adequate renal and metabolic function defined as: calculated glomerular filtration rate (eGFR) (Schwartz formula), or radioisotope GFR >=90 milliliters/minutes (mL/min)/1.73 meter square (m^2); or a serum creatinine within the institutional reference range upper limit of normal (for age/gender, if available).
* Adequate liver function defined as: bilirubin (sum of conjugated + unconjugated) <=1.5 x upper limit of normal (ULN) for age, aspartate aminotransaminase (AST) and alanine transaminase (ALT) <=2.5 x ULN; AST/ALT may be <5 x ULN at baseline if disease under treatment involves the liver (requires radiographic confirmation of liver involvement).
* Adequate cardiac function defined as: left ventricular ejection fraction (LVEF) of either >=50% by ECHO or greater than institutional lower limit of normal (LLN) by echocardiogram (ECHO) (while not receiving medications for cardiac function), corrected QT using Bazett's (QTcB) interval <450 milliseconds (msecs).

Exclusion Criteria:

* Part 2 ONLY: Previous treatment with dabrafenib, another RAF inhibitor, or a mitogen-activated protein kinase (MEK) inhibitor (exception: prior treatment with sorafenib is permitted).
* Malignancy OTHER than the BRAF mutant malignancy under study.
* Had chemotherapy or radiotherapy within 3 weeks (or 6 weeks for nitrosoureas or mitomycin C) prior to administration of the first dose of study treatment.
* The subject has received an investigational product within the following time period prior to the first dosing day in the current study: 28 days or 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is warranted by the data).
* History of another malignancy. Exception: (a) Subjects who have been successfully treated and are disease-free for 3 years, (b) a history of completely resected non-melanoma skin cancer, (c) successfully treated in situ carcinoma, (d) CLL in stable remission are eligible.
* Current use of a prohibited medication or herbal preparation or requires any of these medications during the study.
* Unresolved toxicity greater than National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0 Grade 2 or higher from previous anti-cancer therapy, including major surgery except those that in the opinion of the investigator are not clinically relevant given the known safety/toxicity profile of dabrafenib (e.g., alopecia and/or peripheral neuropathy related to platinum or vinca alkaloid based chemotherapy).
* Has leukaemia.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dabrafenib and its excipients.
* Autologous or allogeneic stem cell transplant within 3 months prior to enrolment [NOTE: subjects with evidence of active graph versus host disease are excluded].
* History of myocardial infarction, severe or unstable angina, peripheral vascular disease or familial QTc prolongation.
* Subjects with abnormal cardiac valve morphology (>=grade 2) documented by echocardiogram (NOTE: subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study).
* Subjects with moderate valvular thickening.
* Known, uncontrolled cardiac arrhythmias (except sinus arrhythmia) within the past 24 weeks
* Uncontrolled medical conditions (e.g., diabetes mellitus, hypertension, liver disease or uncontrolled infection), psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol; or unwillingness or inability to follow the procedures required in the protocol.
* Presence of active GI disease or other condition (e.g., small bowel or large bowel resection) that will interfere significantly with the absorption of drugs.
* Hepatitis B Virus, or Hepatitis C Virus infection (subjects with laboratory evidence of Hepatitis B Virus clearance may be enrolled).
* Pregnant females as determined by positive human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* Lactating females who are actively breast feeding.

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2013-05-23 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (25):
- United States (8):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Seattle, Washington
- Novartis Investigative Site, Parkville, Victoria, Australia
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Copenhagen, Denmark
- France (4):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (3):
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Berlin
- Israel (2):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
- Novartis Investigative Site, Milan, Italy
- Spain (2):
  - Novartis Investigative Site, Esplugues de Llobregat. Barcelona
  - Novartis Investigative Site, Madrid
- United Kingdom (2):
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Whitlock JA, Geoerger B, Dunkel IJ, Roughton M, Choi J, Osterloh L, Russo M, Hargrave D. Dabrafenib, alone or in combination with trametinib, in BRAF V600-mutated pediatric Langerhans cell histiocytosis. Blood Adv. 2023 Aug 8;7(15):3806-3815. doi: 10.1182/bloodadvances.2022008414. PMID 36884302
- [Derived] Hargrave DR, Bouffet E, Tabori U, Broniscer A, Cohen KJ, Hansford JR, Geoerger B, Hingorani P, Dunkel IJ, Russo MW, Tseng L, Dasgupta K, Gasal E, Whitlock JA, Kieran MW. Efficacy and Safety of Dabrafenib in Pediatric Patients with BRAF V600 Mutation-Positive Relapsed or Refractory Low-Grade Glioma: Results from a Phase I/IIa Study. Clin Cancer Res. 2019 Dec 15;25(24):7303-7311. doi: 10.1158/1078-0432.CCR-19-2177. PMID 31811016
- [Derived] Kieran MW, Geoerger B, Dunkel IJ, Broniscer A, Hargrave D, Hingorani P, Aerts I, Bertozzi AI, Cohen KJ, Hummel TR, Shen V, Bouffet E, Pratilas CA, Pearson ADJ, Tseng L, Nebot N, Green S, Russo MW, Whitlock JA. A Phase I and Pharmacokinetic Study of Oral Dabrafenib in Children and Adolescent Patients with Recurrent or Refractory BRAF V600 Mutation-Positive Solid Tumors. Clin Cancer Res. 2019 Dec 15;25(24):7294-7302. doi: 10.1158/1078-0432.CCR-17-3572. Epub 2019 Sep 10. PMID 31506385
- [Derived] Wang J, Yao Z, Jonsson P, Allen AN, Qin ACR, Uddin S, Dunkel IJ, Petriccione M, Manova K, Haque S, Rosenblum MK, Pisapia DJ, Rosen N, Taylor BS, Pratilas CA. A Secondary Mutation in BRAF Confers Resistance to RAF Inhibition in a BRAFV600E-Mutant Brain Tumor. Cancer Discov. 2018 Sep;8(9):1130-1141. doi: 10.1158/2159-8290.CD-17-1263. Epub 2018 Jun 7. PMID 29880583

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 19 centers in eight participating countries: Australia (1), Canada (1), Denmark (1), Germany (1), France (4), Spain (1), United Kingdom (2), and United States (8).
Pre-assignment Details: Patients participated in only either Part 1 (Dose Escalation) or Part 2 (Tumor specific expansion) of the study.
Groups:
- Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg); Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg); Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg); Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg): Repeat dose, dose escalation study in patients with any BRAF V600 mutation-positive solid tumor using a modified Rolling 6 Design (RSD). The RSD was built on the classic 3+3 design, but allowed for continued recruitment of subjects while the data from the first 3 subjects in each cohort was collected (up to 6 subjects per cohort). The starting dose was 3 mg/kg with subsequent dose levels: 3.75 mg/kg, 4.5 mg/kg, 5.25 mg/kg and 6.0 mg/kg.
- Part 2 (Tumor Specific Expansion): Cohort 1 Low-Grade Gliomas (LGG): Subjects with low-grade gliomas with BRAF V600 mutations will receive the single selected final dose (based on MTD and the age of the subjects) from Part 1 on Day 1. Repeat dosing will begin from Day 2, twice daily till end of study.
- Part 2 (Tumor Specific Expansion): Cohort 2 High-Grade Gliomas (HGG): Subjects with high-grade gliomas with BRAF V600 mutations will receive the single selected final dose (based on MTD and the age of the subjects) from Part 1 on Day 1. Repeat dosing will begin from Day 2, twice daily till end of study.
- Part 2 (Tumor Specific Expansion): Cohort 3 Langerhans Cell Histiocytosis (LCH): Subjects with LCH with BRAF V600 mutations will receive the single selected final dose (based on MTD and the age of the subjects) from Part 1 on Day 1. Repeat dosing will begin from Day 2, twice daily till end of study.
- Part 2 (Tumor Specific Expansion): Cohort 4 Miscellaneous Tumors (Other): Subjects with other tumors with BRAF V600 mutations will receive the single selected final dose (based on MTD and the age of the subjects) from Part 1 on Day 1. Repeat dosing will begin from Day 2, twice daily till end of study.
Period: Overall Study
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) | Part 2 (Tumor Specific Expansion): Cohort 1 Low-Grade Gliomas (LGG) | Part 2 (Tumor Specific Expansion): Cohort 2 High-Grade Gliomas (HGG) | Part 2 (Tumor Specific Expansion): Cohort 3 Langerhans Cell Histiocytosis (LCH) | Part 2 (Tumor Specific Expansion): Cohort 4 Miscellaneous Tumors (Other)
Started (All subjects who received at least one dose of study treatment were included in All treated population and Safety population) | 3 | 10 | 8 | 6 | 17 | 28 | 11 | 2
DLT Evaluable Population (Part 1 subjects fulfilling the All Treated population criteria, and having received an adequate treatment for the first 28 days to enable an appropriate evaluation of study drug related DLTs) | 3 | 10 | 8 | 6 | 0 | 0 | 0 | 0
PK Population (Subjects fulfilling the All Treated population criteria and for whom pharmacokinetic sample(s) were obtained and analyzed) | 3 | 10 | 8 | 6 | 17 | 28 | 11 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 10 | 8 | 6 | 17 | 28 | 11 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 7 | 5 | 4 | 11 | 20 | 4 | 2
Not completed — Enrolled in a rollover study | 0 | 3 | 2 | 1 | 6 | 6 | 7 | 0
Not completed — Progressive disease | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) | Part 2 (Tumor Specific Expansion): Cohort 1 Low-Grade Gliomas (LGG) | Part 2 (Tumor Specific Expansion): Cohort 2 High-Grade Gliomas (HGG) | Part 2 (Tumor Specific Expansion): Cohort 3 Langerhans Cell Histiocytosis (LCH) | Part 2 (Tumor Specific Expansion): Cohort 4 Miscellaneous Tumors (Other) | Total
Number analyzed (Participants) | 3 | 10 | 8 | 6 | 17 | 28 | 11 | 2 | 85
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.33 (5.132) | 11.30 (5.355) | 6.58 (5.445) | 7.17 (3.189) | 9.65 (5.195) | 12.32 (3.692) | 5.52 (3.390) | 9.50 (10.607) | 9.46 (5.051)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 3 | 3 | 8 | 11 | 4 | 0 | 35
  Male | 2 | 5 | 5 | 3 | 9 | 17 | 7 | 2 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 0 | 2 | 3 | 0 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 4
  White | 3 | 8 | 7 | 6 | 13 | 22 | 11 | 2 | 72
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events (AEs) in Part 1 (Dose Escalation)
Description: The distribution of adverse events was done via the analysis of frequencies for treatment emergent Adverse Events, Serious Adverse Events and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters. Only descriptive analysis performed.
Time Frame: From study treatment start date till 28 days safety follow-up, assessed up to approximately 90 months
Population: Safety population. Deaths occurring more than 28 days after the last dose of study drug were not included in the on-treatment deaths. All deaths included on-treatment deaths and those occurring more than 28 days after the last dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg)
Number analyzed (Participants) | 3 | 10 | 8 | 6
Participants
  All deaths | 0 | 0 | 0 | 1
  On-treatment deaths | 0 | 0 | 0 | 1
  Adverse Events (AEs) | 3 | 10 | 8 | 6
  AEs suspected to be drug related | 3 | 10 | 8 | 5
  Serious Adverse Events (SAEs) | 0 | 5 | 5 | 3
  SAEs suspected to be drug related | 0 | 2 | 2 | 1
  Fatal SAEs | 0 | 0 | 0 | 1
  Fatal SAEs suspected to be drug related | 0 | 0 | 0 | 0
  AEs leading to discontinuation | 0 | 0 | 1 | 0
  AEs requiring dose interruptions | 1 | 5 | 6 | 5
  AEs requiring dose reductions | 0 | 2 | 3 | 1
  AEs requiring dose reductions or interruptions | 1 | 5 | 6 | 5

2. Primary Outcome: Maximum Concentration (Cmax) of Dabrafenib
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. Cmax of dabrafenib was listed and summarized using descriptive statistics.
Time Frame: Week 1 Day 1, Week 3 Day 15
Population: Pharmacokinetic population. Only participants with an evaluable PK sample collected at each timepoint were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 4,5 mg/kg: All patients at recommended dose phase 2 (RP2D) of 4,5 mg/kg in Part 2 study cohorts (Cohort 1 Low-Grade Gliomas (LGG), Cohort 2 High-Grade Gliomas (HGG), Cohort 3 Langerhans cell histiocytosis (LCH) and Cohort 4 Miscellaneous tumors including melanoma and papillary thyroid carcinoma (Other)) were pooled together.
- Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 5.25 mg/kg: All patients at recommended dose phase 2 (RP2D) of 5.25 mg/kg in Part 2 study cohorts (Cohort 1 Low-Grade Gliomas (LGG), Cohort 2 High-Grade Gliomas (HGG), Cohort 3 Langerhans cell histiocytosis (LCH) and Cohort 4 Miscellaneous tumors including melanoma and papillary thyroid carcinoma (Other)) were pooled together.
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 4,5 mg/kg | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 5.25 mg/kg
Number analyzed (Participants) | 3 | 10 | 8 | 6 | 27 | 31
ng/mL
  Week 1 Day 1: number analyzed (Participants) | 2 | 10 | 8 | 6 | 27 | 31
  Week 1 Day 1 | 1820 (38.0) | 1250 (61.5) | 1250 (529.9) | 1900 (45.0) | 1340 (82.6) | 1550 (56.8)
  Week 3 Day 15: number analyzed (Participants) | 3 | 10 | 8 | 6 | 26 | 29
  Week 3 Day 15 | 1470 (37.7) | 1260 (48.1) | 1580 (49.2) | 1710 (56.4) | 1450 (57.8) | 1310 (49.4)

3. Primary Outcome: Area Under the Concentration-time Curve Over the Dosing Interval (AUC(0-τ)) and AUC From Zero to Infinity (AUC(0-inf)) of Dabrafenib
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. AUC(0-τ) and AUC(0-inf) of dabrafenib were to be listed and summarized using descriptive statistics.
Time Frame: Week 1 Day 1
Population: Pharmacokinetic population. Due to limited dabrafenib PK data collected for Day 1 (up to 4 hours post-dose PK data only), no reliable AUC(0-t) and AUC (0-inf) PK parameters were collected/calculated.
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 4,5 mg/kg | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 5.25 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Pre-dose (Trough) Concentration (C Tau) of Dabrafenib and Its Metabolites
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. Pre-dose (trough) concentration (C tau) was to be listed and summarized using descriptive statistics for dabrafenib and its metabolites (hydroxy-dabrafenib [GSK2285403], carboxy-dabrafenib [GSK2298683], and desmethyl-dabrafenib [GSK2167542]).
Time Frame: Week 3 Day 15
Population: Pharmacokinetic population. For each parameter, only participants with an evaluable PK sample collected were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 4,5 mg/kg | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 5.25 mg/kg
Number analyzed (Participants) | 3 | 10 | 8 | 6 | 26 | 29
ng/mL
  dabrafenib | 11.9 (276.5) | 39.8 (176.1) | 50.7 (121.0) | 11.0 (67.5) | 42.7 (135.9) | 22.8 (209.5)
  hydroxy-dabrafenib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  carboxy-dabrafenib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  desmethyl-dabrafenib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: The AUC(0-t) of Dabrafenib Metabolites
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. Area under the time-concentration curve from time zero (pre-dose) to last time of quantifiable concentration (AUC[0-t]) dabrafenib metabolites (hydroxy-dabrafenib [GSK2285403], carboxy-dabrafenib [GSK2298683], and desmethyl-dabrafenib [GSK2167542]) were to be listed and summarized using descriptive statistics.
Time Frame: Week 1 Day 1, Week 3 Day 15
Population: Pharmacokinetic population. Due to limited dabrafenib PK data collected for Day 1 (up to 4 hours post-dose PK data only), no reliable AUC(0-t) PK parameters were collected/calculated.
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 4,5 mg/kg | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 5.25 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: The AUC(0-tau) of Dabrafenib and Its Metabolites
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. Area under the time-concentration curve from time zero (pre-dose) to last time of quantifiable concentration (AUC(0-tau) of dabrafenib and its metabolites (hydroxy-dabrafenib [GSK2285403], carboxy-dabrafenib [GSK2298683], and desmethyl-dabrafenib [GSK2167542]) were to be listed and summarized using descriptive statistics.
Time Frame: Week 1 Day 1, Week 3 Day 15
Population: Pharmacokinetic population. Due to limited dabrafenib PK data collected for Day 1 (up to 4 hours post-dose PK data only), no reliable AUC(0-tau) PK parameters were collected/calculated.
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 4,5 mg/kg | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 5.25 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Apparent Total Clearance of the Drug From Plasma After Oral Administration (CL/F) of Dabrafenib
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. CL/F of dabrafenib was to be listed and summarized using descriptive statistics.
Time Frame: Week 1 Day 1, Week 3 Day 15
Population: Pharmacokinetic population. Due to limited dabrafenib PK data collected for Day 1 (up to 4 hours post-dose PK data only), no reliable CL/F PK parameters were collected/calculated.
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 4,5 mg/kg | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 5.25 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Maximum Concentration (Cmax) of Dabrafenib Metabolites
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. Cmax of dabrafenib metabolites (hydroxy-dabrafenib [GSK2285403], carboxy-dabrafenib [GSK2298683], and desmethyl-dabrafenib [GSK2167542]) were listed and summarized using descriptive statistics.
Time Frame: Week 1 Day 1, Week 3 Day 15
Population: Pharmacokinetic population. For each parameter, only participants with an evaluable PK sample collected at each timepoint were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 4,5 mg/kg | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 5.25 mg/kg
Number analyzed (Participants) | 3 | 10 | 8 | 6 | 27 | 31
ng/mL
  hydroxy-dabrafenib @ Week 1 Day 1: number analyzed (Participants) | 2 | 10 | 8 | 6 | 26 | 31
  hydroxy-dabrafenib @ Week 1 Day 1 | 811 (24.7) | 662 (66.7) | 473 (1643.7) | 1370 (43.9) | 694 (77.9) | 894 (58.2)
  hydroxy-dabrafenib @ Week 3 Day 15: number analyzed (Participants) | 3 | 10 | 8 | 6 | 26 | 29
  hydroxy-dabrafenib @ Week 3 Day 15 | 673 (62.8) | 726 (37.6) | 752 (32.8) | 1010 (51.5) | 772 (50.1) | 711 (43.4)
  carboxy-dabrafenib @ Week 1 Day 1: number analyzed (Participants) | 2 | 10 | 7 | 6 | 27 | 31
  carboxy-dabrafenib @ Week 1 Day 1 | 1720 (90.6) | 1300 (55.7) | 824 (291.3) | 4250 (67.0) | 1650 (161.2) | 2330 (97.6)
  carboxy-dabrafenib @ Week 3 Day 15: number analyzed (Participants) | 3 | 10 | 8 | 6 | 26 | 29
  carboxy-dabrafenib @ Week 3 Day 15 | 4700 (51.7) | 6410 (28.0) | 9650 (35.9) | 11200 (28.4) | 8280 (45.9) | 7970 (30.0)
  desmethyl-dabrafenib @ Week 1 Day 1: number analyzed (Participants) | 2 | 10 | 6 | 6 | 21 | 27
  desmethyl-dabrafenib @ Week 1 Day 1 | 13.0 (27.3) | 6.55 (80.5) | 15.4 (103.9) | 23.7 (53.8) | 10.7 (159.4) | 10.1 (88.7)
  desmethyl-dabrafenib @ Week 3 Day 15: number analyzed (Participants) | 3 | 10 | 8 | 6 | 24 | 29
  desmethyl-dabrafenib @ Week 3 Day 15 | 194 (219.4) | 311 (78.9) | 317 (324.9) | 238 (45.6) | 328 (38.8) | 274 (77.4)

9. Secondary Outcome: Time to Reach Maximum (Peak) Plasma Concentration Following Drug Administration (Tmax) of Dabrafenib and Its Metabolites
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. Tmax was listed and summarized using descriptive statistics for dabrafenib and its metabolites (hydroxy-dabrafenib [GSK2285403], carboxy-dabrafenib [GSK2298683], and desmethyl-dabrafenib [GSK2167542]).
Time Frame: Week 1 Day 1, Week 3 Day 15
Population: as for outcome 8
Measure: Median (Full Range); unit: Hour (hr)
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 4,5 mg/kg | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 5.25 mg/kg
Number analyzed (Participants) | 3 | 10 | 8 | 6 | 27 | 31
Hour (hr)
  dabrafenib @ Week 1 Day 1: number analyzed (Participants) | 2 | 10 | 8 | 6 | 27 | 31
  dabrafenib @ Week 1 Day 1 | 2.00 [2.00 to 2.00] | 2.00 [2.00 to 4.00] | 2.00 [0.50 to 4.00] | 2.00 [2.00 to 4.00] | 2.00 [0.50 to 4.00] | 2.00 [0.50 to 4.00]
  dabrafenib @ Week 3 Day 15: number analyzed (Participants) | 3 | 10 | 8 | 6 | 26 | 29
  dabrafenib @ Week 3 Day 15 | 1.00 [1.00 to 2.00] | 2.00 [0.50 to 4.00] | 2.00 [1.00 to 3.00] | 2.00 [1.00 to 3.00] | 2.00 [1.00 to 6.00] | 2.00 [1.00 to 4.00]
  hydroxy-dabrafenib @ Week 1 Day 1: number analyzed (Participants) | 2 | 10 | 8 | 6 | 26 | 31
  hydroxy-dabrafenib @ Week 1 Day 1 | 4.00 [4.00 to 4.00] | 4.00 [2.00 to 4.00] | 3.00 [0.50 to 4.00] | 3.00 [2.00 to 4.00] | 4.00 [2.00 to 4.00] | 4.00 [2.00 to 4.00]
  hydroxy-dabrafenib @ Week 3 Day 15: number analyzed (Participants) | 3 | 10 | 8 | 6 | 26 | 29
  hydroxy-dabrafenib @ Week 3 Day 15 | 2.00 [1.00 to 3.00] | 2.50 [1.00 to 4.00] | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 3.00] | 2.00 [1.00 to 6.00] | 2.00 [1.00 to 4.00]
  carboxy-dabrafenib @ Week 1 Day 1: number analyzed (Participants) | 2 | 10 | 7 | 6 | 27 | 31
  carboxy-dabrafenib @ Week 1 Day 1 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00] | 4.00 [0.50 to 4.00] | 4.00 [4.00 to 4.00]
  carboxy-dabrafenib @ Week 3 Day 15: number analyzed (Participants) | 3 | 10 | 8 | 6 | 26 | 29
  carboxy-dabrafenib @ Week 3 Day 15 | 6.00 [4.00 to 8.00] | 4.00 [3.00 to 8.00] | 4.00 [3.00 to 8.00] | 4.00 [3.00 to 4.00] | 4.00 [0.00 to 8.00] | 4.00 [2.00 to 8.00]
  desmethyl-dabrafenib @ Week 1 Day 1: number analyzed (Participants) | 2 | 10 | 6 | 6 | 21 | 27
  desmethyl-dabrafenib @ Week 1 Day 1 | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00] | 4.00 [0.50 to 4.00] | 4.00 [4.00 to 4.00]
  desmethyl-dabrafenib @ Week 3 Day 15: number analyzed (Participants) | 3 | 10 | 8 | 6 | 24 | 29
  desmethyl-dabrafenib @ Week 3 Day 15 | 2.00 [0.00 to 8.00] | 2.00 [0.50 to 8.00] | 1.50 [0.00 to 8.00] | 1.50 [0.00 to 3.00] | 2.00 [0.00 to 8.00] | 1.00 [0.00 to 8.00]

10. Secondary Outcome: Elimination Half Life (T½) of Dabrafenib and Its Metabolites
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. T1/2 of dabrafenib and its metabolites (hydroxy-dabrafenib [GSK2285403], carboxy-dabrafenib [GSK2298683], and desmethyl-dabrafenib [GSK2167542]) was listed and summarized using descriptive statistics.
Time Frame: Week 3 Day 15
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hour (hr)
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 4,5 mg/kg | Part 2 (Tumor Specific Expansion): All Patients at Recommended Dose Phase 2 (RP2D) of 5.25 mg/kg
Number analyzed (Participants) | 3 | 10 | 8 | 6 | 25 | 29
Hour (hr)
  dabrafenib | 1.98 (0.687) | 2.85 (1.58) | 2.74 (0.840) | 1.56 (0.359) | 3.03 (2.27) | 2.54 (2.44)
  hydroxy-dabrafenib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  carboxy-dabrafenib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  desmethyl-dabrafenib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Incidence of Treatment Emergent Adverse Events (AEs) in Part 2 (Tumor Specific Expansion)
Description: The distribution of adverse events was done via the analysis of frequencies for treatment emergent Adverse Events, Serious Adverse Event and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Time Frame: From study treatment start date till 28 days safety follow-up, assessed up to approximately 90 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 (Tumor Specific Expansion): Cohort 1 Low-Grade Gliomas (LGG) | Part 2 (Tumor Specific Expansion): Cohort 2 High-Grade Gliomas (HGG) | Part 2 (Tumor Specific Expansion): Cohort 3 Langerhans Cell Histiocytosis (LCH) | Part 2 (Tumor Specific Expansion): Cohort 4 Miscellaneous Tumors (Other)
Number analyzed (Participants) | 17 | 28 | 11 | 2
Participants
  All deaths | 0 | 1 | 0 | 0
  On-treatment deaths | 0 | 0 | 0 | 0
  Adverse Events (AEs) | 17 | 26 | 11 | 2
  AEs suspected to be drug related | 16 | 26 | 11 | 0
  Serious Adverse Events (SAEs) | 7 | 13 | 6 | 0
  SAEs suspected to be drug related | 1 | 3 | 2 | 0
  Fatal SAEs | 0 | 1 | 0 | 0
  Fatal SAEs suspected to be drug related | 0 | 0 | 0 | 0
  AEs leading to discontinuation | 2 | 1 | 1 | 0
  AEs requiring dose interruptions | 10 | 13 | 7 | 2
  AEs requiring dose reductions | 2 | 4 | 2 | 1
  AEs requiring dose reductions or interruptions | 10 | 13 | 7 | 2

12. Secondary Outcome: Best Overall Response Based on Investigator Assessment Per Response Assessment in Neuro-Oncology (RANO) Criteria for Low Grade Glioma (LLG) Subjects
Description: Overall Response Rate (ORR) was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR).based on Response Assessment in Neuro-Oncology (RANO) criteria for Low Grade Glioma (LLG) and High Grade Glioma (HGG) subjects.
Time Frame: Up to 6 months
Population: All treated population
Measure: Count of Participants; unit: Participants
Groups:
- All LGG Subjects at Recommended Phase 2 Dose (RP2D): All LGG patients who have been assigned to Recommended Phase II Dose (RP2D) across Part 1 and Part 2.
- All LGG Subjects: All LGG subjects in the study
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) | Part 2 (Tumor Specific Expansion): Cohort 1 Low-Grade Gliomas (LGG) | All LGG Subjects at Recommended Phase 2 Dose (RP2D) | All LGG Subjects
Number analyzed (Participants) | 4 | 6 | 6 | 17 | 24 | 33
Participants | 3 | 5 | 4 | 12 | 17 | 24

13. Secondary Outcome: Best Overall Response Based on Investigator Assessment Per Response Assessment in Neuro-Oncology (RANO) Criteria for High Grade Glioma (HGG) Subjects
Description: as for outcome 12
Time Frame: Up to 6 months
Population: All treated population
Measure: Count of Participants; unit: Participants
Groups:
- All HGG Subjects at Recommended Phase 2 Dose (RP2D): All HGG patients who have been assigned to Recommended Phase II Dose (RP2D) across Part 1 and Part 2.
- All HGG Subjects: All HGG subjects in the study
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 2 (Tumor Specific Expansion): Cohort 2 High-Grade Gliomas (HGG) | All HGG Subjects at Recommended Phase 2 Dose (RP2D) | All HGG Subjects
Number analyzed (Participants) | 3 | 4 | 28 | 28 | 35
Participants | 2 | 1 | 7 | 7 | 10

14. Secondary Outcome: Effect of Weight on Total Apparent Clearance (CL/F) of Dabrafenib Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of Dabrafenib can be described using a two-compartment model with a delayed 1st order absorption (Alag1, Ka) and an inducible elimination (CL/F) that consists of a base clearance (constant over time, CL0/F) and a dose- and time-dependent inducible clearance (CLind/F). The PopPK analysis examined the influence of demographics (i.e., weight) on the pharmacokinetics of dabrafenib. The effect of weight on total apparent clearance (CL/F) of dabrafenib estimated with the PopPK model is summarized in this record.
Time Frame: Day 1-Predose, 0.5, 2 and 4 hours post dose; Day 15-Predose, 0, 0.5, 1, 2, 3, 4, 6 and 8 hours post dose.
Population: All subjects who received at least one dose of dabrafenib in Part 1 and 2 and provided an evaluable PK profile. All trametinib and dabrafenib concentration-time data were combined and included in a population PK analysis that examined the influence of demographics on the PK of study treatment.
Measure: Number; unit: coefficient
Groups:
- Part 1 and Part 2 - All Participants With PK Data: Participants in the study (all doses and all tumor types) with available pharmacokinetic data
Arm/Group | Part 1 and Part 2 - All Participants With PK Data
Number analyzed (Participants) | 85
coefficient | 0.223

15. Secondary Outcome: Effect of Weight on Volume of Distribution (V/F) of Dabrafenib Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of Dabrafenib can be described using a two-compartment model with a delayed 1st order absorption (Alag1, Ka) and an inducible elimination (CL/F) that consists of a base clearance (constant over time, CL0/F) and a dose- and time-dependent inducible clearance (CLind/F). The PopPK analysis examined the influence of demographics (i.e., weight) on the pharmacokinetics of dabrafenib. The effect of weight on volume of distribution (V/F) of dabrafenib estimated with the PopPK model is summarized in this record.
Time Frame: Day 1-Predose, 0.5, 2 and 4 hours post dose; Day 15-Predose, 0, 0.5, 1, 2, 3, 4, 6 and 8 hours post dose.
Population: as for outcome 14
Measure: Number; unit: coefficient
Arm/Group | Part 1 and Part 2 - All Participants With PK Data
Number analyzed (Participants) | 85
coefficient | 0.593

16. Secondary Outcome: Effect of Weight on Absorption Rate (ka) of Dabrafenib Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of Dabrafenib can be described using a two-compartment model with a delayed 1st order absorption (Alag1, Ka) and an inducible elimination (CL/F) that consists of a base clearance (constant over time, CL0/F) and a dose- and time-dependent inducible clearance (CLind/F). The PopPK analysis examined the influence of demographics (i.e., weight) on the pharmacokinetics of dabrafenib. The effect of weight on absorption rate (ka) of dabrafenib estimated with a PopPK model is summarized in this record.
Time Frame: Day 1-Predose, 0.5, 2 and 4 hours post dose; Day 15-Predose, 0, 0.5, 1, 2, 3, 4, 6 and 8 hours post dose.
Population: All subjects who received at least one dose of dabrafenib in Part 1 and 2 and provided an evaluable PK profile. The covariate weight did not meet the pre-specified criteria to be considered a significant covariate on Ka based on the goodness-of-fit plots and the decrease of the objective function provided by the PopPK software (NONMEM). Therefore, effect of weight on Ka could not be calculated.
Measure: Number; unit: coefficient
Arm/Group | Part 1 and Part 2 - All Participants With PK Data
Number analyzed (Participants) | 85
coefficient | NA — N/A: covariate weight did not meet the pre-specified criteria required to calculate a result in the PopPK model

17. Secondary Outcome: Effect of Weight on Coefficients for Significant Covariates of Dabrafenib Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of Dabrafenib can be described using a two-compartment model with a delayed 1st order absorption (Alag1, Ka) and an inducible elimination (CL/F) that consists of a base clearance (constant over time, CL0/F) and a dose- and time-dependent inducible clearance (CLind/F). The PopPK analysis examined the influence of demographics (i.e., weight) on the pharmacokinetics of dabrafenib. The effect of weight on coefficients for significant covariates of dabrafenib estimated with a PopPK model is summarized in this record.
Time Frame: Day 1-Predose, 0.5, 2 and 4 hours post dose; Day 15-Predose, 0, 0.5, 1, 2, 3, 4, 6 and 8 hours post dose.
Population: All subjects who received at least one dose of dabrafenib in Part 1 and 2 and provided an evaluable PK profile. The covariate weight did not meet the pre-specified criteria to be considered a significant covariate based on the goodness-of-fit plots and the decrease of the objective function provided by the PopPK software (NONMEM). Therefore, effect of weight on coefficients for significant covariates of dabrafenib could not be calculated.
Measure: Number; unit: coefficient
Arm/Group | Part 1 and Part 2 - All Participants With PK Data
Number analyzed (Participants) | 85
coefficient | NA — N/A: covariate weight did not meet the pre-specified criteria required to calculate a result in the PopPK model

18. Post Hoc Outcome: All Collected Deaths in Parts I and II
Description: On treatment deaths were collected from FPFT up to 28 days after study drug discontinuation, for a maximum duration of 360 weeks in Part I (treatment duration ranged from 5.6 to 356.0 weeks) and a maximum duration of 300 weeks in Part II (treatment duration ranged from 0.3 to 296.0 weeks).
  Deaths post treatment survival follow up were collected after the on- treatment period, up to approximately 7 years. Patients who didn't die during the on-treatment period and had not stopped study participation at the time of data cut-off (end of study) were censored.
Time Frame: up to 360 weeks (on-treatment in Part I), up to 300 weeks (on-treatment in Part II), up to approximately 7 years (study duration)
Population: Clinical database population; all treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) | Part 2 (Tumor Specific Expansion): Cohort 1 Low-Grade Gliomas (LGG) | Part 2 (Tumor Specific Expansion): Cohort 2 High-Grade Gliomas (HGG) | Part 2 (Tumor Specific Expansion): Cohort 3 Langerhans Cell Histiocytosis (LCH) | Part 2 (Tumor Specific Expansion): Cohort 4 Miscellaneous Tumors (Other)
Number analyzed (Participants) | 3 | 10 | 8 | 6 | 17 | 28 | 11 | 2
Participants
  On-treatment deaths | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Post-treatment deaths | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  All deaths | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from First Patient First Treatment (FPFT) up to 28 days after study drug discontinuation, for a maximum duration of 360 weeks in Part I (treatment duration ranged from 5.6 to 356.0 weeks) and a maximum duration of 300 weeks in Part II (treatment duration ranged from 0.3 to 296.0 weeks).
Description: Any sign or symptom that occurs during the treatment period plus 28 days post-treatment.
Arm/Group | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) | Part 2 (Tumor Specific Expansion): Cohort 1 Low-Grade Gliomas (LGG) | Part 2 (Tumor Specific Expansion): Cohort 2 High-Grade Gliomas (HGG) | Part 2 (Tumor Specific Expansion): Cohort 3 Langerhans Cell Histiocytosis (LCH) | Part 2 (Tumor Specific Expansion): Cohort 4 Miscellaneous Tumors (Other)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/10 | 0/8 | 1/6 | 0/17 | 0/28 | 0/11 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 5/10 | 5/8 | 3/6 | 7/17 | 13/28 | 6/11 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 10/10 | 8/8 | 6/6 | 17/17 | 26/28 | 11/11 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) (N=3) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) (N=10) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) (N=8) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) (N=6) | Part 2 (Tumor Specific Expansion): Cohort 1 Low-Grade Gliomas (LGG) (N=17) | Part 2 (Tumor Specific Expansion): Cohort 2 High-Grade Gliomas (HGG) (N=28) | Part 2 (Tumor Specific Expansion): Cohort 3 Langerhans Cell Histiocytosis (LCH) (N=11) | Part 2 (Tumor Specific Expansion): Cohort 4 Miscellaneous Tumors (Other) (N=2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 1 | 1 | 4 | 5 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Corynebacterium infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Salmonellosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stroke-like migraine attacks after radiation therapy (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood culture positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epstein-Barr virus associated lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meningeal disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (Dose Escalation): Dabrafenib Treatment (3 mg/kg) (N=3) | Part 1 (Dose Escalation): Dabrafenib Treatment (3.75 mg/kg) (N=10) | Part 1 (Dose Escalation): Dabrafenib Treatment (4.5 mg/kg) (N=8) | Part 1 (Dose Escalation): Dabrafenib Treatment (5.25 mg/kg) (N=6) | Part 2 (Tumor Specific Expansion): Cohort 1 Low-Grade Gliomas (LGG) (N=17) | Part 2 (Tumor Specific Expansion): Cohort 2 High-Grade Gliomas (HGG) (N=28) | Part 2 (Tumor Specific Expansion): Cohort 3 Langerhans Cell Histiocytosis (LCH) (N=11) | Part 2 (Tumor Specific Expansion): Cohort 4 Miscellaneous Tumors (Other) (N=2)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 3 | 5 | 4 | 3 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0
Monocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 1 | 0 | 3 | 1 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0
Tricuspid valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0
Precocious puberty (Endocrine disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dark circles under eyes (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypermetropia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Papilloedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Periorbital swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retinal exudates (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scleral disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vernal keratoconjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 1 | 2 | 4 | 3 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 0
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cheilosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 3 | 1 | 0 | 2 | 4 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 4 | 3 | 6 | 4 | 4 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 5 | 2 | 2 | 2 | 7 | 4 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Oral mucosal eruption (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 5 | 5 | 4 | 6 | 10 | 9 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 0 | 6 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Catheter site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0
Complication associated with device (General disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 6 | 2 | 3 | 6 | 11 | 3 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 5 | 7 | 5 | 11 | 10 | 4 | 2
Xerosis (General disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 2 | 4 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 1
Enterobiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enterovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 2 | 0 | 1 | 2 | 2 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 1 | 3 | 2 | 1 | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pertussis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Pitted keratolysis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Pustule (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 2 | 2 | 2 | 4 | 3 | 1
Rhinovirus infection (Infections and infestations) | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Skin bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheostomy infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 5 | 2 | 0 | 4 | 4 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 4 | 0 | 1 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0
Viral rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulval abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 1 | 1 | 0 | 2 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 2 | 1 | 0 | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 4 | 2 | 1 | 3 | 0 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 3 | 2 | 0 | 2 | 3 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase decreased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0
Blood bilirubin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood chloride increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 2 | 3 | 5 | 5 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood luteinising hormone increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood prolactin abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood urea decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Carbon dioxide decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Creatinine urine decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 2 | 2 | 2 | 3 | 2 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0
Platelet count decreased (Investigations) | 1 | 2 | 3 | 1 | 1 | 1 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Protein total increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Red blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Respiratory rate decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine albumin/creatinine ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urine protein/creatinine ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 2 | 1 | 1 | 2 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 2 | 2 | 3 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 1 | 2 | 2 | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 3 | 4 | 1 | 6 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 3 | 1 | 3 | 3 | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0 | 1 | 0 | 2 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 0 | 3 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 2 | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 3 | 1 | 1 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 3 | 2 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 3 | 4 | 3 | 3 | 4 | 5 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2 | 2 | 4 | 4 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1 | 1 | 3 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ligament pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2 | 2 | 3 | 4 | 3 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lip neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2 | 2 | 3 | 8 | 4 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 1 | 0 | 2 | 1 | 0
Xanthogranuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 2 | 1 | 2 | 2 | 1 | 0
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dysmetria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 8 | 3 | 2 | 8 | 10 | 4 | 0
Hemianopia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oculofacial paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Periodic limb movement disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 4 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Anger (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 2 | 1 | 1 | 1 | 3 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Dysphemia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Emotional disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Middle insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Haemoglobinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 4 | 1 | 3 | 4 | 1 | 0
Renal tubular disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 4 | 3 | 3 | 8 | 6 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 0
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1 | 2 | 1 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 2 | 0 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 3 | 3 | 4 | 3 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 1 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 2 | 3 | 3 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 0
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 4 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 6 | 3 | 4 | 7 | 9 | 5 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2 | 2 | 1 | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ephelides (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 1 | 0 | 2 | 3 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 2 | 1 | 3 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 2 | 4 | 4 | 3 | 0
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 | 2 | 0 | 4 | 0 | 0
Lentigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail pigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 2 | 5 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 4 | 2 | 3 | 6 | 8 | 3 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 | 1 | 5 | 3 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 0 | 2 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 1 | 3 | 0 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 4 | 1 | 1 | 0
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 3 | 3 | 1 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Steroid therapy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 1 | 2 | 2 | 4 | 1 | 0
Hypotension (Vascular disorders) | 1 | 1 | 2 | 0 | 1 | 0 | 3 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT01677741/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT01677741/SAP_001.pdf